CLINICAL TRIAL: NCT03726099
Title: Efficacy and Safety of 14-day Concomitant Therapy for Helicobacter Pylori: A Pilot Study
Brief Title: Efficacy and Safety of 14-day Concomitant Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018SDU-QILU-G004
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Concomitant Therapy; Rescue treatment
MeSH Terms: interventions — Esomeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14d concomitant therapy (Experimental): Patients will receive a 14-day concomitant therapy containing esomeprazole, amoxicillin, tetracycline and furazolidone.
  Interventions: Drug: esomeprazole, amoxicillin, furazolidone，tetracycline

INTERVENTIONS:
Drug: esomeprazole, amoxicillin, furazolidone，tetracycline — Patients will go through a gastroscopy and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day concomitant therapy containing esomeprazole 40mg bid, amoxicillin 1000mg bid , furazolidone 100mg bid and tetracycline 500mg qid.

SUMMARY:
The purpose of this study is to evaluate efficacy of a 14-day concomitant therapy for the third-line treatment of Helicobacter pylori infection, and whether it is safe while maintaining an ideal eradication rates.

DETAILED DESCRIPTION:
Helicobacter pylori infects half of the world's population. H.pylori eradication is an effective approach to reduce the risk of developing gastric cancer. However, eradication rates of first-line therapy decreased over years due to the rapidly increasing antibiotic resistance of H. pylori worldwide. An ideal rescue therapeutic regimen to cure refractory H.pylori infection is currently warranted. Few published paper evaluated the efficacy of 14-day furazolidone containing concomitant therapy in the third line treatment. This study aims to propose a new concomitant therapy for the patients with two or more treatment failure, and then evaluates whether adverse effects are tolerable. .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with persistent H. pylori infection.
* Patients failed at least three different standard eradication therapies before. Previous standard eradication therapy was defined as a 10-day or 14-day quadruple regimen designed according to Maastricht V report.

Exclusion Criteria:

* Patients unable or unwilling to receive gastroscopy.
* Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastorectomy, acute GI bleeding and advanced gastric cancer.
* History of allergy to any of the drugs used in the study.
* Severe concomitant cardiovascular, respiratory, or endocrine diseases, clinically significant renal or hepatic disease, hematologic disorders and any other clinically significant medical condition that could increase risk.
* Currently pregnant or lactating.
* Severe neurologic or psychiatric disorders.
* Alcohol abuse or drug addiction.
* Patients with compliance lower than 90% in any previous treatment are not included.
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rates | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infection. The ITT analysis includes all the patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of adverse events happening | 6 months
  Common adverse events will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) during the treatment process.
Changes of dyspepsia symptoms after Helicobacter pylori eradication | 6 months
  A list of dyspepsia symptoms will be recorded. Difference of dyspepsia symptoms before and after the therapy will be compared.
The rate of good compliance | 6 months
  Patients taken over 90% of drugs are considered to have a good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China